CLINICAL TRIAL: NCT02519231
Title: A Multi-Center, Double-Blinded, Randomized, Phase IV 6-Month Pilot Study to Compare Bleeding Patterns, Satisfaction and Quality of Life Among New Copper 380A IUD Users Treated With Naproxen Sodium (440mg Twice Daily) Versus Placebo
Brief Title: Copper IUD Treatment Observation Study
Acronym: CITROS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Cook County Hospital (Other); Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Emily Godfrey, Associate Professor of Family Medicine and OB/GYN, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000323
Record Dates: First submitted 2015-06-05; First posted 2015-08-10 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Menorrhagia
Keywords: IUD; naproxen; bleeding
MeSH Terms: conditions — Menorrhagia; Hemorrhage | interventions — Naproxen; Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): This study arm includes naproxen as potential treatment for heavy or prolonged bleeding or dysmenorrhea may provide useful preliminary data for a larger, adequately powered placebo-controlled comparative trial testing additional promising treatments, such as tranexamic acid.
  Interventions: Drug: Naproxen
- placebo (Placebo Comparator): This study arm includes capsules that are exactly like the active treatment medication (naproxen), but there is no active treatment medication in these tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Naproxen 440mg 1x pid
  Other Names: Intervention
  Arms: Treatment
Drug: Placebo — Placebo tablet 440mg 1x pid
  Other Names: Control
  Arms: placebo

SUMMARY:
Studies indicate that bleeding irregularities and dysmenorrhea are common reasons for copper IUD method discontinuation. Some evidence suggests that non-steroidal anti-inflammatory medications (NSAIDs) can help improve bleeding during Cu-IUD use. However, these studies did not examine NSAID use with the TCu380A specifically, nor did they evaluate readily available NSAIDs such as over-the-counter naproxen. For this reason, the investigators propose a pilot trial in which new TCu380A users complaining of heavy or prolonged menstrual bleeding or spotting after 1 month of use are randomized to naproxen or placebo to be taken the first 7 days of menstruation for three consecutive cycles, and then observed for one cycle without treatment.

DETAILED DESCRIPTION:
The Copper IUD (Cu-IUD) is the most widely used IUD in the world, and its use in the United States (US) is on the rise. The Cu-IUD is considered one of the most effective contraception methods, being as effective as permanent sterilization but having the convenience of being reversible should a woman decide to conceive.2 The Copper 380A (TCu380A) is the only Cu-IUD available in the US; of all Cu-IUDs, the TCu380A is considered the most effective. Despite its increasing popularity in the US, studies indicate that bleeding irregularities and dysmenorrhea are common reasons for method discontinuation. Some evidence suggests that non-steroidal anti-inflammatory medications (NSAIDs) can help improve bleeding during Cu-IUD use. However, these studies did not examine NSAID use with the TCu380A specifically, nor did they evaluate readily available NSAIDs such as over-the-counter naproxen. For this reason, the investigators propose a pilot trial in which new TCu380A users complaining of heavy or prolonged menstrual bleeding or spotting after 1 month of use are randomized to naproxen or placebo to be taken the first 7 days of menstruation for three consecutive cycles, and then observed for one cycle without treatment. The number of bleeding/spotting days will be compared using Student t-test. In addition to assessing how well naproxen reduces incidence and amount of bleeding, the investigators will also assess the use of naproxen and TCu380A on quality of life, sexual function, method satisfaction, menstrual pain, and adverse events. By measuring these variables, the investigators will assess both positive and negative consequences of TCu380A use, ensuring that harm does not outweigh benefits.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 and < 49 years. We are including a wide range of ages because women of all ages request TCu380A. While we recognize that some women approaching menopause (median age = 51.4 years) may have changes in their baseline menstruation, we trust that clinicians enrolling the patients into the study will ensure that these women meet all inclusion (i.e., regular cycles) and exclusion criteria (i.e., do not have diagnosis of menorrhagia).

  * Requesting to have TCu380A IUD inserted as contraceptive method.
  * English-speaking.
  * Regular menstrual cycles ranging 21-35 days apart.
  * Generally healthy.
  * Willing to attend a 4- to 6-week follow-up visit and complete surveys.

Exclusion Criteria:

* Known or suspected pregnancy.

  * Contraindications to NSAID use. This includes underlying heart failure, chronic renal disease, chronic liver disease, peptic ulcer disease, or history of upper gastrointestinal bleed, and allergy to NSAIDs.
  * Current regular use of a NSAID.
  * Unwilling to avoid use of NSAIDs (except for study medication) for the duration of the study.
  * Current diagnosis of menorrhagia, metrorrhagia, symptomatic uterine fibroids, or endometrial polyps.
  * Use of depot medroxyprogesterone acetate (DMPA) or levonorgestrel-releasing intrauterine device (LNG IUD) within the previous 3 months.
  * Postpartum in the past 4 weeks. The average day in which non-breastfeeding postpartum women ovulate is 25 days after birth, indicating that menstrual cycles can resume after the 4th postpartum week.
  * Existing medical condition for which placement of TCu380A IUD is a contraindication according to the Centers for Disease Control and Prevention Medical Eligibility Criteria (MEC 4 medical conditions; see Appendix A).
  * Currently breastfeeding.
  * Previous use of the TCu380A.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Godfrey, MD,MPH, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Harborview Medical Center, Seattle, Washington
  - UW Neighborhood Clinic Northgate, Seattle, Washington
  - Hall Health Center, Seattle, Washington
  - University of Washington Medical Centers, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All datasets used and analysed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Until 12/2022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2016 to May 2017, 34 women enrolled into the study, of whom 28 were randomized.
Pre-assignment Details: Subjects who completed the baseline questionnaires were contacted 4-5 weeks later to determine eligibility for randomization to a treatment arm. Participants were eligible to be randomized if they reported any change in menstrual bleeding since their TuC380A insertion, were willing to forgo NSAIDs, and willing to record their daily bleeding.
Groups:
- Treatment: This study arm includes naproxen as potential treatment for heavy or prolonged bleeding or dysmenorrhea may provide useful preliminary data for a larger, adequately powered placebo-controlled comparative trial .
  Naproxen: Naproxen 440mg 1x bid for fist 7 days of menstrual cycle
- Placebo: This study arm includes capsules that are exactly like the active treatment medication (naproxen), but there is no active treatment medication in these tablets.
  Placebo: Placebo tablet 440mg 1x bid for first 7 days of menstruation
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 14 | 14
Completed | 12 (One was lost to follow up and never took the treatment. another never turned in bleeding diary.) | 8 (Six participants never turned in their bleeding diaries.)
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were no significant differences of baseline characteristics between the groups. The majority participating in the study had a mean age of 29 years, were white, had Bachelor's degree or higher, married/living with their partner and nulliparous.
Groups:
- Treatment: This study arm includes naproxen as potential treatment for heavy or prolonged bleeding or dysmenorrhea may provide useful preliminary data for a larger, adequately powered placebo-controlled comparative trial testing additional promising treatments, such as tranexamic acid.
  Naproxen: Naproxen 440mg 1x bid
- Placebo: This study arm includes capsules that are exactly like the active treatment medication (naproxen), but there is no active treatment medication in these tablets.
  Placebo: Placebo tablet 1x bid
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [23 to 35] | 29.3 [21 to 42] | 29.3 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Days of Bleeding and Spotting, Spotting Only and Bleeding Only for the 84 Day Treatment Cycles and Last 28 Day Post-treatment Cycle
Description: Number of bleeding and spotting, spotting only and bleeding only days given as mean. We calculated the mean difference and 95% confidence interval between the two treatment groups and provided the p-value of means.
Time Frame: 4 months
Population: Population who submitted bleeding diaries at the end of the 6-month trial. We used intention-to-treat and included all data we had. We excluded missing data
Measure: Mean (Standard Error); unit: days
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 8
days
  Bleeding or spotting days first 84 days | 29.2 (4.5) | 23.0 (2.8)
  Bleeding or spotting days last 28 days | 9.3 (1.9) | 9.6 (0.9)
  Bleeding only days first 84 days | 15.7 (2.1) | 15.5 (1.8)
  Bleeding only days last 28 days | 4.8 (1.0) | 6.6 (1.2)
  Spotting only days first 84 days | 13.5 (5.1) | 7.5 (1.7)
  Spotting only days last 28 days | 4.5 (2.0) | 3.0 (0.8)
Statistical Analysis 1: Comparison: Treatment vs Placebo; We originally planned to enroll 60 subjects based on other similar studies that evaluated treatment for bleeding among women using contraception; as reported by Cohen et al., a sample size of 42 provided 80% power to detect a difference of 7 bleeding/spotting days in 30 days by two-sample t-test, allowing for an expected 20% drop-out; Test type: Superiority; p = .11, t-test, 2 sided — The threshold for statistical significance was p =0.05; For days with bleeding/spotting outcomes, we used independent t-tests to compare the unadjusted mean difference between groups; Mean Difference (Net) = -1.76, Standard Error of Mean 5 — Treatment Difference = Naproxen - Placebo; We designed the study to include another site, in addition to the UW site enrolled participants. After 6 months of failed active recruitment at the other site, we discontinued that site from the study. Resources did not permit us to contract with an alternative recruitment site, and thus the protocol was revised to enroll 32 participants at the Seattle site only

2. Secondary Outcome: Percentage Reporting Moderate-heavy/Heavy Menses, Often/Always Menstrual Cramping and 7 or More Days of Menstrual Bleeding for the 84-day Treatment Months and 28-day Post-treatment Month
Description: Percentage reporting moderate-heavy/heavy menses, often/always menstrual cramping and 7 or more days of menstrual bleeding during the first 84 days and the last 28 days. We also report % difference and p-value between the two treatment groups.
Time Frame: 4 months
Population: Includes participants who responded to the monthly questionnaires, based on intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 13 | 14
Participants
  Month 1 : Moderate heavy or heavy bleeding | 7 | 7
  Month 1 : Menstrual bleeding length 7+ days | 8 | 5
  Month 1 : Often/always cramping | 1 | 5
  Month 1 : Unexpected bleeding | 6 | 5
  Month 2 : Moderate heavy or heavy bleeding | 4 | 8
  Month 2 : Menstrual bleeding length 7+ days | 8 | 5
  Month 2 : Often/always cramping | 1 | 1
  Month 2 : Unexpected bleeding | 7 | 7
  Month 3 : Moderate heavy or heavy bleeding | 6 | 7
  Month 3 : Menstrual bleeding length 7+ days | 6 | 5
  Month 3 : Often/always cramping | 1 | 1
  Month 3 : Unexpected bleeding | 1 | 5
  Month 4 : Moderate heavy or heavy bleeding | 7 | 5
  Month 4 : Menstrual bleeding length 7+ days | 6 | 6
  Month 4 : Often/always cramping | 3 | 1
  Month 4 : Unexpected bleeding | 5 | 6
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 4 months
Description: Daily diary asked patients to complete side effects while in study
Groups:
- Placebo: This study arm includes capsules that are exactly like the active treatment medication (naproxen), but there is no active treatment medication in these tablets.
  Placebo: Placebo tablet 440mg 1x bid
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
(1) Small sample size, which did not provide sufficient power to detect differences between the groups; (2) Missing bleeding diaries of 40% of placebo users and 15% of naproxen users. Our findings should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. If requested in writing, Institution and Investigator will withhold such Public Presentation for up to an additional ninety (90) days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02519231/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT02519231/ICF_001.pdf